CLINICAL TRIAL: NCT03511027
Title: Next-generation Medication Dispenser to Improve Care at Home for Community-dwelling Elderly
Brief Title: Medication Dispenser to Improve Care at Home for the Elderly
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Lee Verweel (Other)
Collaborators: CapitalCare Group Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Lee Verweel, Manager, West Park Healthcare Centre, West Park Healthcare Centre
Organization: West Park Healthcare Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I2P2: AceAge
Record Dates: First submitted 2018-03-23; First posted 2018-04-27 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Medication Adherence; Cognitive Impairment
Keywords: Medication Adherence; Medication Dispensing; Homecare; Elderly
MeSH Terms: conditions — Medication Adherence; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This study will utilize a multi-site randomized controlled trial design. One week prior to discharge from inpatient rehab, consenting patients will be randomly assigned to receive medication self-management education only (SME) or medication self-management education + Karie (SME+K).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (SME + Karie Device) (Experimental): Patients randomly assigned to receive SME+Karie will 1) undergo Screening for Self Medication Readiness to determine self-management capacity, 2) will receive self-medication education (SME) by a study Occupational Therapist, and 3) receive a 5-day self-medication performance assessment by an Registered Nurse prior to discharge. In addition, this group will receive orientation to the Karie Automated Medication Delivery by the study Occupational Therapist. The participants in the intervention arm will use the Karie device for all applicable medications for the study duration.
  Interventions: Device: SME + Karie Device
- Control (SME only) (Active Comparator): West Park has a "Self-Medication Education Program" policy in place which seeks to establish independent medication self-medication capacity during the inpatient stay. Eligibility criteria for SME include a need to manage medications independently at home; stabilized on medication (as per pharmacist/physician discretion); and mild-moderate cognitive/physical impairments (as per an OT assessment). During SME participants receive training by an Occupational Therapist, followed by a 5-day self-medication performance assessment by an Registered Nurse prior to discharge. Participants in the SME group will fill prescriptions as usual for the duration of study.
  Interventions: Other: SME only

INTERVENTIONS:
Device: SME + Karie Device — For the duration of the study, participants will use the Karie device to promote medication adherence. The Karie device prompts users to take their medication in the right amount at the right time.
  Arms: Intervention (SME + Karie Device)
Other: SME only — At discharge, participants will be provided with self-medication education.
  Arms: Control (SME only)

SUMMARY:
The purpose of this study is to investigate the efficacy of the Karie Automated Medication delivery device in enhancing medication adherence among a group of elderly patients with mild to moderate cognitive decline.

DETAILED DESCRIPTION:
Given the risks associated with poor adherence and the apparent contribution of good adherence to reducing hospitalizations and emergency department (ED) visits, interventions for promoting good adherence should be pursued. To this end, a number of devices have been developed to promote medication adherence, though with limited success due to reliability, cost, etc. The purpose of this study is to investigate the efficacy of the Karie Automated Medication Delivery Device in enhancing medication adherence among a group of community-dwelling patients immediately following discharge from inpatient rehabilitation.

This study will utilize a multi-site randomized controlled trial design. One week prior to discharge from inpatient rehab, consenting patients will be randomly assigned to receive medication self-management education only (SME) or medication self-management education + Karie (SME+K). Both sites (West Park Healthcare Centre, and CapitalCare) will recruit 150 participants for the study. At each site, 75 patients will be in the intervention group (SME + Karie) and 75 will be in the control group (SME only).

ELIGIBILITY:
Inclusion Criteria:

* Need to manage medications independently at home
* Stabilized on medication, as per pharmacist/physician discretion; and
* Mild-moderate cognitive/physical impairments, as per OT assessment
* Montreal Cognitive Assessment (MoCA) score not less than 16
* English speaking

Exclusion Criteria:

* Absent from community for more than one month during study
* Inability to access study site pharmacy following discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Medication Adherence | Baseline (Time 0 Months), 3-months post-baseline(Time 3 Months), 6 months post-baseline (Time 6 Months)
  The Medication Adherence Questionnaire (MAQ) and medication 7 day recall will measure participants adherence to their medications over time.Both of these measures will be taken at the same time-points throughout the study.

SECONDARY OUTCOMES:
Beliefs about medication | Baseline (Time 0M)
  The Beliefs About Medication questionnaire, assesses participants cognitive representations of medication.
Change in Self-Medication Behaviours | Baseline (Time 0M), 3-months post-baseline(Time 3M), 6 months post-baseline (Time 6M)
  The investigators will use the Self-Efficacy for Appropriate Medication Scale (SEAMS) to determine participants behaviours and attitudes about self-medication
Change in Quality of Life | Baseline (Time 0M), 3-months post-baseline(Time 3M), 6 months post-baseline (Time 6M)
  The investigators will use the EQ-5D to measure changes in quality of life throughout the study.
Economic Analysis | 3 months post-baseline (Time 3M), 6 months post-baseline (Time 6M)
  To determine the affect that the Karie device has on economic indicators, the investigators will be observing staffing hours (OT, Pharmacist), medication costs, and medication wastage. This will be documented by staff and will be self-reported.
Change in Healthcare Consumption | Baseline (Time 0M), 3-months post-baseline(Time 3M), 6 months post-baseline (Time 6M)
  To determine any changes in healthcare consumption, the investigators will be observing the number of hospitalizations, visits to the GP, and visits to ER for all causes in all of the participants.
Sociodemographic Factors | Baseline (Time 0M)
  The investigators will be collecting sociodemographic factors such as: Age, Gender, Education, Income, Postal Code.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Pauley, MSc, Principal Investigator — West Park Healthcare Centre

IPD SHARING:
Plan to Share IPD: No
No, individual patient data will only be available to the study investigators identified on the Research Ethics Board applications at each study site.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT03511027/Prot_SAP_000.pdf